CLINICAL TRIAL: NCT06959732
Title: Efficacy and Safety of Zanubrutinib Combined With G-CVP Regimen in Previously Untreated Follicular Lymphoma
Brief Title: Zanubrutinib Combined With G-CVP in Previously Untreated FL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhitao Ying, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/548-4828
Record Dates: First submitted 2025-04-25; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Follicular Lymphoma ( FL)
Keywords: Follicular Lymphoma ( FL); Zanubrutinib; Obinutuzumab; CVP
MeSH Terms: conditions — Lymphoma, Follicular | interventions — zanubrutinib; obinutuzumab; COP protocol 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZG- CVP (Experimental): Zanubrutinib , obinutuzumab , cyclophosphamide , vincristine, and prednisone tablets were used every 21 days as a treatment cycle. Six cycles of treatment were completed, and the efficacy was reviewed every two cycles. Patients with progressive disease (PD) were excluded from the group. MRD was detected after six cycles. If MRD was negative, routine maintenance therapy was performed . If MRD was positive, Zanubrutinib was added to the conventional maintenance therapy for 12 months.
  Interventions: Drug: zanubrutinib, obinutuzumab,combined with CVP

INTERVENTIONS:
Drug: zanubrutinib, obinutuzumab,combined with CVP — Zanubrutinib (160 mg, twice daily [bid]), obinutuzumab (1000 mg on cycle 1 [C1], days 1, 8, and 15; on cycle 2 - 6 [C 2-6], day 1), cyclophosphamide (750 mg/㎡ on day 1), vincristine (1.4 mg/㎡, maximum dose 2 mg on day 1), and prednisone tablets (40 mg/㎡ once daily [qd] orally on days 1-5) were used every 21 days as a treatment cycle. Six cycles of treatment were completed, and the efficacy was reviewed every two cycles. Patients with PD were excluded from the group. MRD was detected after six cycles. If MRD was negative, routine maintenance therapy was performed (obinutuzumab 1000 mg once every 8 weeks, a total of 12 times). If MRD was positive, Zanubrutinib (160 mg, continuous bid) was added to the conventional maintenance therapy for 12 months.

SUMMARY:
The goal of this clinical trial is to learn the efficacy and safety of zanubrutinib in combination with G-CVP in previously untreated follicular lymphoma patients The main questions it aims to answer are: (1) Efficacy and safety of patients receiving zanubrutinib, obinutuzumab combined with cyclophosphamide, vincristine, and prednisone (CVP) regimen. (2) The difference in efficacy of patients with different minimal residual disease (MRD) status after treatment.

Participants will receive zanubrutinib combined with G-CVP, maintenance therapy will be determined by the MRD status after treatment.

DETAILED DESCRIPTION:
Follicular lymphoma (FL), accounting for nearly 20% of non - Hodgkin lymphomas, is an indolent B - cell neoplasm originating from follicular center B cells. Over 90% of patients are at stage Ⅲ/Ⅳ at onset. For stage Ⅲ/Ⅳ patients requiring treatment, CD20 monoclonal antibody - chemotherapy combinations are the most commonly used treatment both domestically and internationally. Though FL has a high response rate to traditional immunochemotherapy, it remains incurable by such means. Also, cytotoxic therapy's side effects are a key concern. There's an urgent need in clinical practice to enhance therapeutic efficacy while reducing side effects.

Obinutuzumab, a type II anti - CD20 monoclonal antibody, stands out from type I by boosting antitumor activity through enhanced direct cytotoxicity (DCD) and antibody - dependent cellular cytotoxicity (ADCC), and cutting complement - dependent cytotoxicity (CDC) - related resistance. Studies comparing obinutuzumab - chemotherapy with rituximab - chemotherapy in untreated FL have confirmed that the former brings sustained progression - free survival (PFS) benefits. Compared to CHOP or bendamustine combinations, it has a lower incidence of grade 3 - 5 adverse events when used with CVP, showing better tolerability. Zanubrutinib, a novel, highly - selective small - molecule BTK inhibitor developed in China, offers superior efficacy and safety due to its high kinase selectivity. Its combination with obinutuzumab has achieved remarkable results in relapsed/refractory FL patients.

In this study, we will treat untreated FL patients with zanubrutinib, obinutuzumab, and CVP chemotherapy. We expect this multi - mechanism drug combination to improve efficacy. Also, by replacing CHOP's anthracycline component, the regimen may provide better safety, thus offering a more effective and safer individualized treatment for untreated FL patients.

Untreated FL patients in the study will receive zanubrutinib, obinutuzumab, and CVP chemotherapy. Then, based on their MRD status, they'll undergo maintenance with either obinutuzumab alone or the combination. The primary endpoint is the complete remission (CR) rate; secondary endpoints include overall response rate (ORR), PFS, overall survival (OS), and adverse event (AE) rates.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible:

1. Histologically confirmed CD20-positive FL (grades 1, 2, or 3a), diagnosed according to the WHO 2022 criteria; 2, Clear indication for treatment: symptoms affecting normal work and life; end-organ dysfunction; cytopenia due to bone marrow involvement by lymphoma; bulky disease (per GELF criteria); persistent or rapidly progressive disease; 3. No prior systemic therapy for lymphoma; 4. Age 18-80 years; 5. Eastern cooperative oncology group (ECOG) performance status (PS) < 2; 6. Expected survival > 2 years; 7. At least one measurable lesion with a longest diameter ≥ 1.5 cm or extranodal lesion ≥ 1 cm; 8. Willingness to participate in the study and comply with treatment and follow-up.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Pregnant or breastfeeding women;
2. Abnormal liver or kidney function, defined as: serum direct/indirect bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), or serum creatinine > 2 × upper limit of normal (ULN); creatinine clearance < 60 mL/min (unless due to lymphoma involvement);
3. History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months;
4. Absolute neutrophil count (ANC) < 1.5 × 10⁹/L, platelets < 75 × 10⁹/L, or hemoglobin < 70 g/L (unless due to bone marrow involvement by lymphoma);
5. Long-term use of strong or moderate CYP3A inducers;
6. Known hypersensitivity to any component of the study drug;
7. Other active malignancies, except: cured non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, superficial bladder cancer, ductal carcinoma in situ, or other malignancies with disease-free survival > 5 years;
8. Severe concurrent infections;
9. Drug abuse, medical, psychological, or social conditions that may interfere with study participation or result evaluation;
10. Investigator-deemed ineligibility for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
CRR | From date of enrollment until the date of first documented CR assessed up to 2.5 years.
  CRR (%) is defined as the number of patients achieving a complete response as a proportion of total patients evaluable for response.

SECONDARY OUTCOMES:
ORR | From date of enrollment until the date of first documented response assessed up to 2.5 years.
  ORR (%) is defined as the number of patients achieving a complete response or partial response as a proportion of total patients evaluable for response.
PFS | From date of enrollment until the date of first documented progression assessed up to 5 years.
  PFS is defined as the time interval from the time of enrollment on this study to the date of PD or death, whichever came first.
OS | From date of enrollment until the date of first documented death assessed up to 5 years.
  OS is defined as the time interval from the time of enrollment in this study to the date of death from any cause. If the subject is alive or the vital status is unknown, OS will be censored at the date that the subject is last known to be alive, or their last contact date.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No